CLINICAL TRIAL: NCT06587061
Title: An Exploratory Clinical Study of HRS-4642 in Combination With Gemcitabine and Albumin-bound Paclitaxel for Neoadjuvant and Adjuvant Treatment of Pancreatic Cancer
Brief Title: HRS-4642 in Combination With AG for Neoadjuvant and Adjuvant Treatment of Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, BAIYONG SHEN, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANC-PERI-IIT-HRS4642-AG
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-4642, Gemcitabine and Albumin-bound Paclitaxel (Experimental): HRS-4642 in Combination With AG for Neoadjuvant and Adjuvant Treatment of Pancreatic Cancer
  Interventions: Drug: HRS-4642+AG

INTERVENTIONS:
Drug: HRS-4642+AG — HRS-4642 in Combination With Gemcitabine and Albumin-bound Paclitaxel will be administrated per dose level in which the patients are assigned.

SUMMARY:
To evaluate the safety and efficacy of HRS-4642 in Combination With AG for Neoadjuvant and Adjuvant Treatment of Pancreatic Cancer

DETAILED DESCRIPTION:
This study is an open, single center, exploratory clinical trial aimed at evaluating the safety and efficacy of HRS-4642 in combination with gemcitabine and albumin-bound paclitaxel for neoadjuvant and adjuvant treatment of pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 and ≤80 years old, male or female;
2. Pathologically or cytologically confirmed ductal adenocarcinoma of the pancreas; and subjects must have at least one measurable lesion as defined by RECIST v1.1;
3. Imaging evaluation met the NCCN guidelines definition of resectable pancreatic cancer (including high-risk resectable) and borderline resectable pancreatic cancer.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
5. Life expectancy ≥ 12 weeks;
6. Adequate marrow and organ function;
7. Female participants of childbearing age must undergo a pregnancy test within one week before the start of the study medication, and the result is negative. They are willing to use a medically recognized and efficient contraceptive method during the study period and within three months after the last administration of the study medication; For male participants whose partners are women of childbearing age, they should agree to use effective methods of contraception during the study period and within 6 months after the last study administration;
8. Patients volunteered to participate in this study and signed informed consent;

Exclusion Criteria:

1. Previously received any anti-tumor therapy;
2. the presence of distant metastatic lesions diagnosed by imaging;
3. Known hypersensitivity to the study drug or any of its components;
4. previous or concurrent other malignant tumors;
5. Participation in a clinical trial of any drug or medical device within 4 weeks prior to the first dose;
6. Received live and attenuated vaccines within 4 weeks prior to the first dose of the investigational drug;
7. previous allogeneic hematopoietic stem cell transplantation or organ transplantation;
8. Patients with severe cardiovascular arterial thromboembolism (e.g., myocardial infarction, unstable angina, stroke), NYHA class 2 or greater cardiac insufficiency, and clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
9. with interstitial lung disease, non-infectious pneumonia or severe and uncontrolled medical illness, acute infections, recent history of major surgery (within 28 days or not yet recovered from side effects);
10. with congenital or acquired immunodeficiencies such as human immunodeficiency virus (HIV) infection, active hepatitis B (positive hepatitis B virus surface antigen [HBsAg] test result at screening together with an HBVDNA test value of ≥10,000 copies/ml [2000 IU/ml]), active hepatitis C (hepatitis C virus antigen [HCV-antibodies] at screening), or active hepatitis C (hepatitis C virus antitoxin [HCV-antibodies] at screening).antibody [HCV-Ab] positive at screening and HCV-RNA positive at the same time), or co-infection with hepatitis B and hepatitis C;
11. Presence of clinically significant acute or chronic pancreatitis; patients at high risk for pancreatitis, e.g., serum amylase and/or lipase concentrations ≥3 times ULN (except when the investigator determines that abnormally elevated amylase and/or lipase are associated with pancreatic cancer);
12. Other situations that the researcher felt should not be included.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | From the first drug administration to within 30 days for the last dose
  AEs are assessed by NCI-CTCAE v5.0
Objective Response Rate (ORR) | Up to approximately 6 months
  Evaluated by RECIST v1.1

SECONDARY OUTCOMES:
Total resection rate | At the time of surgery
  Percentage of subjects who received surgical treatment as a proportion of all subjects
pathologic complete response (pCR) | At the time of surgery
  Number of subjects achieving pCR as a percentage of subjects
R0 resection rate | At the time of surgery
  Number of Subjects Achieving R0 Removal as a Percentage of Subjects
major pathologic response (MPR, CAP Score 0-1) | At the time of surgery
  Number of Subjects Achieving MPR as a Percentage of Subjects
Disease-free survival (DFS) | Up to approximately 6 months
  The time from adjuvant therapy to the occurrence of disease recurrence (local recurrence or distant recurrence) or death from any cause in subjects achieving R0/R1 resection is counted as occurring first
Event-free survival (EFS) | Up to approximately 6 months
  The time from the first dose of neoadjuvant therapy to the occurrence of any event; events include the occurrence of imaging disease progression (based on the date of the imaging test), the occurrence of disease recurrence (local recurrence or distant recurrence) after surgery, and death from any cause, based on the time of the first occurrence
Overall survival (OS) | Up to approximately 12 months
  Time from the date of enrollment to data of death from any cause, or date of lost follow-up, whichever comes first, and otherwise censored at time last known alive.

OTHER OUTCOMES:
CA19-9 response rate | Up to approximately 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China